CLINICAL TRIAL: NCT06069440
Title: Analysis of Kinematical and Muscular Fatigue in Long Distance Swimmers
Brief Title: Kinematical and Muscular Fatigue in Swimmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Luca Puce, Principal Investigator, Universita degli Studi di Genova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DINOGMI-2023
Record Dates: First submitted 2023-09-26; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: muscle fatigue; Neuromuscular Strategy; performance; sEMG; swimming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- swimmers (Experimental)
  Interventions: Other: Swimming Fatigue Task

INTERVENTIONS:
Other: Swimming Fatigue Task — Swim freestyle at a steady, controlled pace until mechanical failure (i.e., inability to maintain the predetermined speed) is reached.

SUMMARY:
During a submaximal task, gradual muscle fatigue occurs, which inevitably results in a decline in performance (mechanical failure). Elite athletes are known to employ unconscious compensatory strategies during fatiguing submaximal tasks in an attempt to delay the onset of mechanical failure as long as possible.

The purpose of this study was to gain valuable insight into the strategies used by elite swimmers to cope with mechanical failure. Twenty-two swimmers were subjected to a swim test consisting of swimming as long as possible at a predetermined and controlled pace. A light strip positioned at the bottom of the pool allows athletes to get feedback on which gait to keep. The kinematics (stroke rate, stroke length, and efficiency index) and electrical activity of 10 muscle groups were analyzed and compared at the beginning of the test (non-fatiguing conditions), just before the athlete lost the ability to maintain the predetermined pace (pre-mechanical failure), and after the athlete lost the ability to maintain the pace (mechanical failure). It is hypothesized that as fatigue becomes more pronounced and the point of inability to maintain a predetermined speed is approached, increased EMG activity will occur in key muscles while other muscle groups may show more obvious signs of fatigue. In addition, changes in the rhythm and coordination of upper limb movements may occur.

ELIGIBILITY:
Inclusion Criteria:

1. Middle- or long-distance swimmer specializing in front crawl
2. At least 3 years of experience in international competition
3. Daily use of flashing light for pace control in aerobic, anaerobic threshold and maximum oxygen consumption training.

Exclusion Criteria:

1) Presence of muscle pain or soreness that could prevent the athlete from performing at their best

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Flexor Carpi Radialis muscle activity | up to 10 minutes
  Electromyographic signal analysis (Root Mean Square)
Biceps Brachii muscle activity | up to 10 minutes
  Electromyographic signal analysis (Root Mean Square)
Triceps Brachii caput lateralis muscle activity | up to 10 minutes
  Electromyographic signal analysis (Root Mean Square)
Deltoideus Lateralis muscle activity | up to 10 minutes
  Electromyographic signal analysis (Root Mean Square)
Latissimus Dorsi muscle activity | up to 10 minutes
  Electromyographic signal analysis (Root Mean Square)
Superior Trapezius muscle activity | up to 10 minutes
  Electromyographic signal analysis (Root Mean Square)
Erector Spinae muscle activity | up to 10 minutes
  Electromyographic signal analysis (Root Mean Square)
Pectoralis Major pars clavicularis muscle activity | up to 10 minutes
  Electromyographic signal analysis (Root Mean Square)
Rectus Femoris muscle activity | up to 10 minutes
  Electromyographic signal analysis (Root Mean Square)
Biceps Femoris muscle activity | up to 10 minutes
  Electromyographic signal analysis (Root Mean Square)
Kinematic parameters | up to 10 minutes
  stroke frequency (time required to complete a stroke cycle)
Kinematic parameters | up to 10 minutes
  stroke length (distance traveled during each stroke cycle))

SECONDARY OUTCOMES:
Flexor Carpi Radialis muscle fatigue | up to 10 minutes
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal
Biceps Brachii muscle fatigue | up to 10 minutes
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal
Triceps Brachii caput lateralis muscle fatigue | up to 10 minutes
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal
Deltoideus Lateralis muscle fatigue | up to 10 minutes
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal
Latissimus Dorsi muscle fatigue | up to 10 minutes
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal
Superior Trapezius muscle fatigue | up to 10 minutes
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal
Erector Spinae muscle fatigue | up to 10 minutes
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal
Pectoralis Major pars clavicularis muscle fatigue | up to 10 minutes
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal
Rectus Femoris muscle fatigue | up to 10 minutes
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal
Biceps Femoris muscle fatigue | up to 10 minutes
  time-course evolution of the median frequency of the power density spectrum (MF [Hz]) of the sEMG signal

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Genova, Genova, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Puce L, Biz C, Ruaro A, Mori F, Bellofiore A, Nicoletti P, Bragazzi NL, Ruggieri P. Analysis of Kinematic and Muscular Fatigue in Long-Distance Swimmers. Life (Basel). 2023 Oct 27;13(11):2129. doi: 10.3390/life13112129. PMID 38004269